CLINICAL TRIAL: NCT02252770
Title: Nitric Oxide Supplementation as a Therapeutic Intervention in Argininosuccinic Aciduria
Brief Title: Nitric Oxide Supplementation in Argininosuccinic Aciduria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sandesh Chakravarthy Sreenath Nagamani, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-33236
Record Dates: First submitted 2014-09-25; First posted 2014-09-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Argininosuccinic Aciduria; Argininosuccinate Lyase Deficiency; Urea Cycle Disorders
Keywords: ASA; ASLD; UCD
MeSH Terms: conditions — Argininosuccinic Aciduria; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitric oxide supplement arm (Active Comparator): During this arm, subjects will receive a lozenge with nitric oxide supplement
  Interventions: Dietary Supplement: Nitric oxide supplement
- Placebo Arm (Placebo Comparator): During this arm, subjects will receive placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nitric oxide supplement — Each active comparator supplement is an all natural nitric oxide supplement. Subjects will take one lozenge twice a day.
  Arms: Nitric oxide supplement arm
Dietary Supplement: Placebo — Placebo will not contain nitric oxide supplement.
  Arms: Placebo Arm

SUMMARY:
This is a study involving a dietary supplement. Patients with argininosuccinic aciduria will be randomly assigned to receive either a nitric oxide dietary supplement or placebo for 2 weeks, and then crossed-over to receive the other treatment for two weeks.

The investigators expect to see that : 1) Patients with ASA will have a decreased ability for their arteries to dilate due to nitric oxide deficiency, 2) Treatment of ASA with the nitric oxide supplement will improve the ability of their arteries to dilate, and 3) Through the testing of subjects' fibroblasts (cells in connective tissue that produce collagen and other fibers), the investigators hope to predict which patients may respond NO supplementation.

DETAILED DESCRIPTION:
The investigators will perform a double blind, randomized, placebo-controlled, crossover study of NO supplementation in ASA patients assessing endothelial function and blood pressure as primary endpoints, and markers of nitric oxide production as exploratory endpoints.

Subjects will receive a nitrite-restricted diet prior to the start and during the trial period. The dietary protein prescriptions will not be altered. After screening, informed consent, subjects will undergo study procedures at the Clinical Research Center (CRC) at Texas Children's Hospital, Houston, TX.

Safety laboratories will be performed. Fibroblast and lymphoblast cultures will be established for subsequent studies.A baseline assessment of the vascular endothelial NO production and function will be assessed using FMD of brachial artery using standard techniques (1). Subjects will be randomized to receive either dietary nitric oxide supplement or placebo for 2 weeks, and then crossed-over to receive the other treatment for two weeks. The Investigational Pharmacy Services at Texas Children's Hospital will assign the initial treatment group randomly in a 1:1 ratio using established randomization procedures. Following randomization, subjects will be receive either Neo40® 40 mg/kg/day in two divided doses) or placebo for 14 days. This dose is the dietary supplemental dose and was well-tolerated in the investigators proof of concept treatment subject as well as other clinical studies in cardiovascular disease. Subjects will return on day 14 to the CRC where they will undergo assessment of FMD of the brachial artery, repeated BP measurements, and assay of NO status. The subjects will then be crossed over to receive the alternative treatment and the study procedures will be repeated in identical fashion to the initial arm.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of ASA based on biochemical, enzymatic, or genetic testing
* Capable of completing study procedures
* History of compliance with diet and treatment

Exclusion Criteria:

* An active infection (viral or bacterial), any condition(s) that may precipitate a metabolic decompensation
* A hypersensitivity to nitrite
* A serum creatinine > 1.5 times above the normal
* A clinical or laboratory abnormality of Grade 3 or greater according to the CTCAE V4.0 (except elevations of AST or ALT which are a part of the disease) which in the view of the Investigator compromises safety

Ages: 8 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial function as assessed by FMD of brachial artery | 2 weeks
  The primary outcome measures will be vascular endothelial function as assessed by the flow mediated dilatation (FMD) of the brachial artery measured by Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh CS Nagamani, MD, FACMG, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Nagamani SC, Campeau PM, Shchelochkov OA, Premkumar MH, Guse K, Brunetti-Pierri N, Chen Y, Sun Q, Tang Y, Palmer D, Reddy AK, Li L, Slesnick TC, Feig DI, Caudle S, Harrison D, Salviati L, Marini JC, Bryan NS, Erez A, Lee B. Nitric-oxide supplementation for treatment of long-term complications in argininosuccinic aciduria. Am J Hum Genet. 2012 May 4;90(5):836-46. doi: 10.1016/j.ajhg.2012.03.018. Epub 2012 Apr 26. PMID 22541557
- [Background] Nagamani SC, Lee B, Erez A. Optimizing therapy for argininosuccinic aciduria. Mol Genet Metab. 2012 Sep;107(1-2):10-4. doi: 10.1016/j.ymgme.2012.07.009. Epub 2012 Jul 20. PMID 22841516
- See also: Sandesh CS Nagamani — http://www.bcm.edu/people/view/b22371a1-ffed-11e2-be68-080027880ca6
- See also: Baylor College of Medicine, Department of Molecular and Human Genetics — http://www.bcm.edu/departments/molecular-and-human-genetics